CLINICAL TRIAL: NCT03851653
Title: Lifestyle Intervention for Obstructive Sleep Apnoea in Adults: A Randomized Controlled Trial
Brief Title: Lifestyle Intervention for OSA in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Almudena Carneiro Barrera, Teaching and Research Academic Staff, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INTERAPNEA-2019
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; weight loss; lifestyle intervention; continuous positive airway pressure; OSA; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Intervention Group (LIG) (Experimental): Participants from this group will receive a cognitive-behavioral intervention addressing weight loss and lifestyle habits such as hypocaloric diet, moderate exercise, smoking and alcohol avoidance, and sleep hygiene. This behavioral intervention will be combined with the usual treatment for OSA, i.e. CPAP.
  Interventions: Behavioral: Lifestyle Intervention
- Control group (No Intervention): Participants from the control group will not receive any type of intervention apart from the usual care (CPAP).

INTERVENTIONS:
Behavioral: Lifestyle Intervention — Cognitive-behavioural intervention for weight loss and lifestyle change
  Arms: Lifestyle Intervention Group (LIG)

SUMMARY:
Obstructive sleep apnoea (OSA) is characterized by the presence in the polysomnogram test of more than five apnoea-hypopnoea episodes per hour of sleep (apnoea-hypopnoea index, AHI > 5), each episode lasting more than 10 seconds and being accompanied by oxygen desaturation or arousal. The prevalence of this syndrome is worryingly high (9% to 38%), affecting more men than women. OSA has an important negative impact on physical/psychological health and on these patient's quality of life. The gold-standard treatment for OSA is the continuous positive airway pressure (CPAP). However, CPAP compliance is really low, this device requiring a continuous chronic use in order to improve OSA and to avoid the relapse. Furthermore, it does not address OSA risk factors such as obesity and unhealthy lifestyle habits. Consequently, non-surgical and non-pharmacological interventions such as weight loss and lifestyle interventions are necessary and recommended by the American Academy of Sleep Medicine (AASM). The objective of this project, therefore, is the development and evaluation of a cognitive-behavioural treatment program for patients with moderate-severe OSA. The treatment will pursued weight loss through hypocaloric diet and moderate exercise, smoking and alcohol avoidance, and sleep hygiene. The efficacy of this treatment will be assessed in comparison with CPAP, in a short and medium term. This intervention could be considered a good alternative/combined management to the usual treatment of OSA (CPAP) once its efficacy to reduce and even cure OSA symptoms is demonstrated, especially if it is still effective in the long-term.

ELIGIBILITY:
Inclusion Criteria:

* Previous clinical diagnosis of moderate/severe OSA (AHI > 15) by a healthcare professional.
* Male patients aged between 18-65 years.
* Body mass index > 25 kg/m2.
* Use of CPAP
* Motivation to participate in the study.
* Signed informed consent form.

Exclusion Criteria:

* Sleep disorder other than OSA
* Clinically significant psychiatric, neurological, or medical disorders other than OSA
* Use of prescription drugs or clinically significant drugs affecting sleep

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Change in apnoea-hypopnoea index (AHI) from baseline to post-intervention. | Post-intervention (2 months)
  Change in apnoea (airflow reduction greater than or equal to 90%) and hypopnoea (airflow reduction greater than or equal to 30%) episodes per hour of sleep, from baseline to post-intervention.

SECONDARY OUTCOMES:
Change in oxygen desaturation index (ODI) from baseline to post-intervention. | Post-intervention (2 months)
  Change in the number of oxygen desaturations greater than or equal to 4%/h from baseline to post-intervention.
Change in oxygen saturation (SaO2) mean from baseline to post-intervention | Post-intervention (2 months)
  Change in the average of oxygen saturation from baseline to post-intervention
Change in oxygen saturation (SaO2) nadir from baseline to post-intervention | Post-intervention (2 months)
  Minimum oxygen saturation from baseline to post-intervention
Change in sleep efficiency from baseline to post-intervention | Post-intervention (2 months)
  Change in the total sleep time/total time in bed from baseline to post-intervention
Change in light sleep (N1 and N2 stages) from baseline to post-intervention | Post-intervention (2 months)
  Change in the percentage of light sleep (N1 and N2 stages) from baseline to post-intervention
Change in deep sleep (N3 stage) from baseline to post-intervention | Post-intervention (2 months)
  Change in the percentage of deep sleep (N3 stage) from baseline to post-intervention
Change in rapid eye movement (REM) sleep from baseline to post-intervention | Post-intervention (2 months)
  Change in the percentage of REM sleep from baseline to post-intervention
Change in apnoea-hypopnoea index (AHI) in REM sleep from baseline to post-intervention. | Post-intervention (2 months)
  Change in apnoea-hypopnoea index (AHI) in REM sleep from baseline to post-intervention.
Change in apnoea-hypopnoea index (AHI) in NREM sleep from baseline to post-intervention. | Post-intervention (2 months)
  Change in apnoea-hypopnoea index (AHI) in NREM sleep from baseline to post-intervention.
Change in excessive daytime sleepiness (EDS) from baseline to post-intervention | Post-intervention (2 months)
  Change in the difficulty in maintaining a desired level of wakefulness, measured by the Epworth sleepiness scale (ESS) from baseline to post-intervention. ESS is a 4-point scale (0 = no chance of dozing, 1 = slight chance of dozing, 2 = moderate chance of dozing, 3 = high chance of dozing) that measures the usual chances of dozing off or falling asleep while engaged in eight different activities. An ESS total score from 0 to 9 is considered to be normal while an ESS total score > 9 indicates high daytime sleepiness.
Change in Pittsburgh Sleep Quality Index (PSQI) from baseline to post-intervention. | Post-intervention (2 months)
  Change in Pittsburgh Sleep Quality Index (PSQI) from baseline to post-intervention. This scale includes a total of 19 self-rated items combined to form seven component scores i.e., subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction), each of which has a range of 0-3 points. The sum of these seven PSQI component scores is considered to obtain a global PSQI score (ranging from 0-21), with higher scores indicating poorer sleep quality.
Change in Wake After Sleep Onset (WASO) from baseline to post-intervention | Post-intervention (2 months)
  Change in Wake After Sleep Onset (WASO; minutes) from baseline to post-intervention
Change in body weight (kg) from baseline to post-intervention | Post-intervention (2 months)
  Change in body weight (kg) from baseline to post-intervention
Change in fat mass (kg) from baseline to post-intervention | Post-intervention (2 months)
  Change in fat mass (kg) from baseline to post-intervention
Change in mean blood pressure (mm HG) from baseline to post-intervention | Post-intervention (2 months)
  Change in mean blood pressure (mm HG) from baseline to post-intervention
Change in plasma glucose (mg/dL) from baseline to post-intervention | Post-intervention (2 months)
  Change in plasma glucose (mg/dL) from baseline to post-intervention
Change in total cholesterol (mg/dL) from baseline to post-intervention | Post-intervention (2 months)
  Change in total cholesterol (mg/dL) from baseline to post-intervention
Change in total triglycerides (mg/dL) from baseline to post-intervention | Post-intervention (2 months)
  Change in total triglycerides (mg/dL) from baseline to post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Gualberto Buela-Casal, PhD, Study Director — Universidad de Granada; Jonatan R. Ruiz, PhD, Study Director — Universidad de Granada; Almudena Carneiro-Barrera, MD, Principal Investigator — Universidad de Granada
Locations (1):
- University of Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie results in a publication
Time Frame: After publication

REFERENCES:
- [Background] Carneiro-Barrera A, Diaz-Roman A, Guillen-Riquelme A, Buela-Casal G. Weight loss and lifestyle interventions for obstructive sleep apnoea in adults: Systematic review and meta-analysis. Obes Rev. 2019 May;20(5):750-762. doi: 10.1111/obr.12824. Epub 2019 Jan 4. PMID 30609450
- [Background] Sanchez AI, Martinez P, Miro E, Bardwell WA, Buela-Casal G. CPAP and behavioral therapies in patients with obstructive sleep apnea: effects on daytime sleepiness, mood, and cognitive function. Sleep Med Rev. 2009 Jun;13(3):223-33. doi: 10.1016/j.smrv.2008.07.002. Epub 2009 Feb 7. PMID 19201228
- [Background] Aiello KD, Caughey WG, Nelluri B, Sharma A, Mookadam F, Mookadam M. Effect of exercise training on sleep apnea: A systematic review and meta-analysis. Respir Med. 2016 Jul;116:85-92. doi: 10.1016/j.rmed.2016.05.015. Epub 2016 May 21. PMID 27296826
- [Background] Iftikhar IH, Bittencourt L, Youngstedt SD, Ayas N, Cistulli P, Schwab R, Durkin MW, Magalang UJ. Comparative efficacy of CPAP, MADs, exercise-training, and dietary weight loss for sleep apnea: a network meta-analysis. Sleep Med. 2017 Feb;30:7-14. doi: 10.1016/j.sleep.2016.06.001. Epub 2016 Jun 28. PMID 28215266
- [Background] Jurado-Gamez B, Guglielmi O, Gude F, Buela-Casal G. Effects of continuous positive airway pressure treatment on cognitive functions in patients with severe obstructive sleep apnoea. Neurologia. 2016 Jun;31(5):311-8. doi: 10.1016/j.nrl.2015.03.002. Epub 2015 May 11. English, Spanish. PMID 25976943
- [Background] Carneiro-Barrera A, Amaro-Gahete FJ, Diaz-Roman A, Guillen-Riquelme A, Jurado-Fasoli L, Saez-Roca G, Martin-Carrasco C, Ruiz JR, Buela-Casal G. Interdisciplinary Weight Loss and Lifestyle Intervention for Obstructive Sleep Apnoea in Adults: Rationale, Design and Methodology of the INTERAPNEA Study. Nutrients. 2019 Sep 15;11(9):2227. doi: 10.3390/nu11092227. PMID 31540168
- [Derived] Vazquez-Lorente H, Herrera-Quintana L, Ruiz JR, Amaro-Gahete FJ, Carneiro-Barrera A. Impact of weight loss and lifestyle intervention on vitamin D in men with obstructive sleep apnea: The INTERAPNEA trial. Sleep Med. 2025 Apr;128:37-45. doi: 10.1016/j.sleep.2025.01.011. Epub 2025 Jan 21. PMID 40023509
- [Derived] Carneiro-Barrera A, Amaro-Gahete FJ, Lucas JF, Saez-Roca G, Martin-Carrasco C, Lavie CJ, Ruiz JR. Weight loss and lifestyle intervention for cardiorespiratory fitness in obstructive sleep apnea: The INTERAPNEA trial. Psychol Sport Exerc. 2024 May;72:102614. doi: 10.1016/j.psychsport.2024.102614. Epub 2024 Feb 17. PMID 38369267
- [Derived] Carneiro-Barrera A, Amaro-Gahete FJ, Saez-Roca G, Martin-Carrasco C, Palmeira AL, Ruiz JR. Interdisciplinary Weight Loss and Lifestyle Intervention for Daily Functioning and Psychiatric Symptoms in Obstructive Sleep Apnea: The INTERAPNEA Randomized Clinical Trial. J Clin Psychiatry. 2023 Jun 12;84(4):22m14502. doi: 10.4088/JCP.22m14502. PMID 37339363
- [Derived] Carneiro-Barrera A, Amaro-Gahete FJ, Jurado-Fasoli L, Saez-Roca G, Martin-Carrasco C, Tinahones FJ, Ruiz JR. Effect of a Weight Loss and Lifestyle Intervention on Dietary Behavior in Men with Obstructive Sleep Apnea: The INTERAPNEA Trial. Nutrients. 2022 Jun 30;14(13):2731. doi: 10.3390/nu14132731. PMID 35807913
- [Derived] Carneiro-Barrera A, Amaro-Gahete FJ, Guillen-Riquelme A, Jurado-Fasoli L, Saez-Roca G, Martin-Carrasco C, Buela-Casal G, Ruiz JR. Effect of an Interdisciplinary Weight Loss and Lifestyle Intervention on Obstructive Sleep Apnea Severity: The INTERAPNEA Randomized Clinical Trial. JAMA Netw Open. 2022 Apr 1;5(4):e228212. doi: 10.1001/jamanetworkopen.2022.8212. PMID 35452108